CLINICAL TRIAL: NCT01385020
Title: Effect of Gemfibrozil on the Safety and Pharmacokinetics of Red Yeast Rice in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201105057MC
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Subjects
Keywords: Red yeast rice; Gemfibrozil; Drug-drug interaction; Pharmacokinetics
MeSH Terms: interventions — Gemfibrozil; red yeast rice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemfibrozil & red yeast rice (LipoCol) (Experimental): The effect of gemfibrozil on the pharmacokinetics of red yeast rice capsule (LipoCol) after administering single-dose combination in healthy subjects
  Interventions: Drug: Gemfibrozil & red yeast rice (LipoCol)

INTERVENTIONS:
Drug: Gemfibrozil & red yeast rice (LipoCol) — The effect of gemfibrozil on the pharmacokinetics of red yeast rice capsule (LipoCol) after administering single-dose combination in healthy subjects.

SUMMARY:
Red yeast rice capsule (LipoCol Forte)is a nature product that has been demonstrated a significant cholesterol lowering effect which might be caused by addictive and/or synergistic effects of lovastatin (monacolin K) with other monacolins and substances in capsules. The usual dose of red yeast rice capsule(LipoCol Forte)for hypercholesterolemia is one capsule twice/day.

Gemfibrozil is a fibric acid derivative (fibrate). It can reduce the levels of triglycerides and increase the levels of high-density lipoprotein cholesterol (HDL-C). Patients with mixed lipid disorders may therefore benefit from a combination of a statin and a fibrate. Although the combination of a fibrate and a statin is highly effective,concerns about an increased incidence of myopathy and even rhabdomyolysis have limited the widespread use of such combinations. Such combination therapies are prone to drug-drug interactions, which can lead to altered pharmacokinetic profiles of either drug, an effect observed for many statins in combination with fibrates. However, the drug-drug interactions have not been reported between red yeast rice capsule and gemfibrozil.

The objective of the study is to evaluate the effect of gemfibrozil on the plasma concentrations of lovastatin and its active form, lovastatin acid, from red yeast rice capsule in healthy volunteers. In addition, the investigators also measure the plasma concentration of creatine kinase (CK) and co-enzyme Q10 for safety assessment.

DETAILED DESCRIPTION:
A randomized,crossover study design with 2 periods was used. The washout time between the periods was 4 days. In first period, 600 mg red yeast rice capsule (LipoCol) was administered orally with 240 mL water at 8 AM. In second period, subjects took 600 mg gemfibrozil (two Lopid 300-mg capsule) at 7 AM and 7 PM for 2 days. On day 3, subjects took 600 mg gemfibrozil at 7 AM then 600 mg red yeast rice capsule was administered orally with 240 mL water at 8 AM. The volunteers had fasted overnight, a breakfast and dinner was severed 0.5 hour after the administration of gemfibrozil. In addition, a high fat breakfast was served 0.5 hour before and standard meal was served 4 and 10 hours after the administration of red yeast rice (LipoCol).

The blood samples will be drawn prior to the dosing, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after the administration of red yeast rice(LipoCol)for detecting the plasma concentration of lovastatin and lovastatin acid. In addition, the blood samples will be drawn prior to the dosing, and 1, 2, 4, 6 and 12 hours after the administration of red yeast rice (LipoCol) for detecting the plasma concentration of creatine kinase (CK) and co-enzyme Q10.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at the age of 20-40 years old and be able to sign informed consent prior to study.
2. Body weight must be above 45 kilograms (kg) and within -20 to +20% of ideal body weight.
3. No clinically significant abnormalities were judged by the principal investigator based on the medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.

Exclusion Criteria:

1. Use of any prescription medication, over-the-counter medications or vitamins within 14 days prior to dosing.
2. Participation in any clinical investigation within 2 months prior to dosing or longer as required by local regulation.
3. Donation or loss of more than 500 milliliter (mL) blood within 3 months prior to dosing.
4. Presence of liver disease (Glutamic Oxaloacetic Transaminase (GOT), Glutamic Pyruvic Transaminase (GPT) or Total-bilirubin greater than 2-fold normal values) or renal disease (blood urea nitrogen (BUN) or creatinine greater than 1.5-fold normal values).
5. Creatine kinase (CK) value greater than 1.5-fold normal value.
6. A known hypersensitivity to statins and fibrates or their analogs.
7. Permanent confinement to an institution.
8. Individuals are judged by the investigator or co-investigator to be undesirable as subjects for other reasons.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacokinetic parameters of lovastatin and lovastatin acid in healthy subjects | 1 week
  Plasma concentrations of lovastatin and lovastatin acid were detected at following time: (Pre-dose (T0), and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours after oral administration red yeast rice capsule (LipoCol) with or without gemfibrozil All pharmacokinetic parameters were determined with lovastatin and lovastatin acid concentrations by non-compartment methods.

SECONDARY OUTCOMES:
Evaluation of the plasma concentration of creatine kinase (CK) and co-enzyme Q10 in healthy subjects | 1 week
  Plasma concentrations of creatine kinase (CK) and co-enzyme Q10 were detected at following time: (Pre-dose (T0), and 1, 2, 4, 6, and 12 hours after oral administration red yeast rice capsule (LipoCol) with or without gemfibrozil)

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan